CLINICAL TRIAL: NCT01767077
Title: Role of Milk Fat Globule Membranes in Dairy Foods: Health Effects in Humans
Acronym: MFGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Lund University (Other); LRF Mjölk, Sweden (Unknown); Arla Foods (Industry); Skånemejerier, Sweden (Unknown); Semper AB, Sweden (Unknown); The Swedish Research Council for Environment, Agricultural Sciences and Spatial Planning (FORMAS) (Other Government); Swedish Nutrition Foundation SNF (Unknown); Vinnova (Other Government); The Swedish Farmers' Foundation for Agricultural Research (Unknown); Livsmedelsföretagen, Sweden (Unknown); Svensk Dagligvaruhandel, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: TvärLivs-MFGM
Record Dates: First submitted 2013-01-09; First posted 2013-01-14 (Estimated); Last update posted 2013-09-25 (Estimated); Status verified 2013-09

CONDITIONS: Hypercholesterolemia
Keywords: Saturated fat; Dairy products; Milk fat globule membrane; Cholesterol; Butter; Cream
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ghee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Butter oil (Placebo Comparator): Daily intake of 40 g butter oil
  Interventions: Dietary Supplement: Butter oil
- Cream (Active Comparator): Daily intake of 100 g cream (40%)
  Interventions: Dietary Supplement: Cream

INTERVENTIONS:
Dietary Supplement: Butter oil — Daily intake of 40 g butter oil
  Arms: Butter oil
Dietary Supplement: Cream — Daily intake of 100 g cream (40%)
  Arms: Cream

SUMMARY:
Investigate the effects of milk fat with or without milk fat globule membranes (MFGM) on blood lipid profile, vascular function, insulin sensitivity, inflammation and gene expression. Overweight subjects will be randomized to one of 2 groups with different types of dairy products: 1)butter oil; 2) cream (milk fat with MFGM).

DETAILED DESCRIPTION:
Dairy foods are a major component of the nordic diet. Epidemiological data suggest potential health effects of dairy foods with regard to obesity related disorders. Low-fat dairy foods have shown to be protective, but also high-fat products have been linked to reduced risk in some studies. It is well known that dairy products increase LDL-cholesterol in blood, but effects on glucose metabolism are unclear. Intervention trials are needed to clarify the health effects of dairy foods. Some data have indicated that cheese and milk may have less hypercholesterolemic effect compared with butter. Our hypothesis is that milk fat globule membranes (MFGM), present in all dairy products except butter, can affect blood lipid profile, vascular function, insulin sensitivity, inflammation and gene expression. Such idea might explain why different dairy products could have different effects on cholesterol levels. The investigators aim to conduct a controlled study to investigate this. Overweight subjects will be randomized to one of 2 groups with different types of dairy products: 1)butter oil; 2) cream (milk fat with MFGM).

ELIGIBILITY:
Inclusion Criteria:

* BMI 25-37
* LDL-cholesterol 2.0-4.5 mmol/l

Exclusion Criteria:

* Use of lipid lowering drugs
* Diagnosed cardiovascular disease or diabetes
* Use of extreme diets
* Food allergies relevant to the study
* Pregnancy or active lactation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterol | 8 weeks

SECONDARY OUTCOMES:
Other major blood lipids | 8 weeks
  HDL-cholesterol, total cholesterol, triglycerides, apolipoproteins
Homeostasis model of assessment - insulin resistance | 8 weeks
  Insulin and glucose
Peripheral blood mononuclear cell gene expression | 8 weeks
Inflammatory markers | 8 weeks
  C-reactive protein, Tumor necrosis factor alfa receptor 2, Interleukin-1-receptor antagonist

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Risérus, Assoc prof, Principal Investigator — Uppsala University
Locations (1):
- Uppsala university, Dept of public health and caring sciences; Clinical nutrition and metabolism, Uppsala, Sweden

REFERENCES:
- [Derived] Rosqvist F, Smedman A, Lindmark-Mansson H, Paulsson M, Petrus P, Straniero S, Rudling M, Dahlman I, Riserus U. Potential role of milk fat globule membrane in modulating plasma lipoproteins, gene expression, and cholesterol metabolism in humans: a randomized study. Am J Clin Nutr. 2015 Jul;102(1):20-30. doi: 10.3945/ajcn.115.107045. Epub 2015 May 27. PMID 26016870